CLINICAL TRIAL: NCT04305964
Title: The Use of Nasal Airway Stent (Nastent®) in Patients With Sleep-disordered Breathing (SDB) Including Snoring and/or Obstructive Sleep Apnea (OSA).
Brief Title: Nasal Airway Stent (Nastent®) Study in OSA
Acronym: Nastent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Prof. Dr. Olivier Vanderveken, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B300201942080
Record Dates: First submitted 2020-03-03; First posted 2020-03-12 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Snoring; Stent
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nastent® users (Experimental): Patients with an established diagnosis of obstructive sleep apnea with apnea/hypopnea-index (AHI) < 20/ hour sleep who receive Nastent® as treatment modality
  Interventions: Device: Nastent® (a distally perforated soft silicon nasal tube); Diagnostic Test: Polygraphy with WatchPAT™ 300

INTERVENTIONS:
Device: Nastent® (a distally perforated soft silicon nasal tube) — Insertion of the Nastent® to nostril during sleep hours
Diagnostic Test: Polygraphy with WatchPAT™ 300 — WatchPAT™ 300 is an innovative diagnostic Home Sleep Apnea Test (HSAT) that utilizes the proprietary Peripheral Arterial Tone signal (PAT™) to enable simple, accurate and reliable sleep apnea testing.
  Other Names: PG

SUMMARY:
This study intends to assess the effect of nasal airway stent (Nasten®) as a treatment modality in patients with sleep-disordered breathing (SDB) including snoring and/or obstructive sleep apnea (OSA). Nastent®, a distally perforated soft silicon nasal tube, is a mechanical splint against collapse of the upper airway at multiple levels. Nastent® might be able to prevent the vibrations caused by fluttering of various parts of the upper airway which leads to snoring. Furthermore, it also potentially secures a patent airway throughout the night securing airflow.

DETAILED DESCRIPTION:
Patients with an established diagnosis of OSA with apnea/hypopnea-index (AHI)< 20/ hour sleep from the ENT department are recruited and informed about the study. After obtaining informed consent and patient inclusion, a baseline portable sleep monitoring at home using WatchPAT™300 for one night is performed. During the next visit the objective size and position of the stent is determined under direct visualization using fiberoptic nasolaryngoscopy. Subsequently, the patients will receive a Nastent® Starter kit (containing 6 different stent sizes of Nastent®, 130, 135, 140, 145, 150 and 155mm) to gradually get accustomed to the stent and to find the right size for them. During the following consultation, a Nastent® classic kit (containing 7 stents of the same size, each can be used for two consecutive nights) is given to the patients to be used for 14 consecutive nights. During the last night of this 14-night period, a follow-up home portable sleep monitoring evaluation using WatchPAT™300 is performed with Nastent® in situ. Afterwards, during the final visit at the outpatient clinic, acceptance of the therapy with Nastent® by the patients is evaluated, and the decision of whether to continue the therapy and to proceed to the purchase of this product as a long-term treatment for the patient or not, is made.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* AHI ≤ 20 per hour of sleep
* Complaints of socially disturbing snoring by the partner of the patient
* Capable of giving informed consent

Exclusion Criteria:

* Craniofacial deformities
* Acute nasal trauma, fracture (during the past 3 months)
* Nasal valve collapse, synechiae and septal perforation, recurrent epistaxis, recent nasopharyngeal surgery, chronic rhinosinusitis with or without polyposis
* Cerebrospinal fluid leaks
* History of past or current psychiatric disorders (psychotic illness, major depression, or acute anxiety attacks as mentioned by the patient), intellectual disability, memory disorders, seizure disorders, neuromuscular disorders, cardiovascular diseases, coagulopathies (thrombocytopenia< 100/µl), lower respiratory tract disorders.
* Pregnancy or willing to become pregnant
* Excessive alcohol or drug use (> 20 alcohol units/week or any use of hard drugs)
* History of sleep medication use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
AHI (apnea-hypopnea index) | At baseline
  Number of apneas and hypopneas per hour of sleep which is an indicator of severity of sleep apnea, (5< normal, 5-15 Mild, 15-30 moderate, <30 severe)
AHI (apnea-hypopnea index) | at follow up after completion of treatment period (an average of three weeks)
  Number of apneas and hypopneas per hour of sleep which is an indicator of severity of sleep apnea, (5< normal, 5-15 Mild, 15-30 moderate, <30 severe)

SECONDARY OUTCOMES:
Epworth sleepiness scale score (ESS) | baseline
  an 8-item questionnaire which takes about three minutes to fill out. It reflects the chance of each person's general level of sleepiness during eight situations of daily life. The subject selects the most appropriate integer score ranging from 0 (would never doze) to 3 (high chance of dozing) for each of the 8 questions. The results are then summed up, with 0 being the minimal and 24 the maximum total ESS score. The higher the ESS score, the higher that person's average sleep propensity in daily life. (0-5=Lower Normal Daytime Sleepiness, 6-10 = Higher Normal Daytime Sleepiness, 11-12 = Mild Excessive Daytime Sleepiness, 13-15 = Moderate Excessive Daytime Sleepiness, 16-24 =Severe Excessive Daytime Sleepiness.)
VAS (visual analogue scale) for snoring | Baseline
  A standard 10-point VAS ranging from 0 (no snoring) to 10 (extreme snoring causing the bed partner to leave the bedroom or sleep separately) will be used to evaluate the subjective status of snoring during sleep. Heavy snoring corresponds to a snoring index of at least 7. A decrease of 3 points after treatment is considered significant. A satisfactory improvements is defined as a reduction to an index that is no longer experiences as bothersome (i.e. <3).
ODI (oxygen desaturation index) | baseline
  The ODI represents the average number of desaturation episodes (≥3%) per hour sleep.
PAT (peripheral arterial tone) signal | baseline
  PAT™ technology is a non-invasive window to the cardiovascular system and autonomic nervous system. Peripheral Arterial Tone (PAT™) signal is a proprietary technology used for non-invasively measuring arterial tone changes in peripheral arterial beds.
Heart rate | baseline
  The number of times a person's heart beats per minute. Normal heart rate range for adults is 60 to 100 beats per minute.
Body position | baseline
  Percentage of supine, prone, left, right, upright position
Snoring | baseline
  Snoring loudness in decibels
Oxygen saturation (SaO2) | baseline
  A measurement of the percentage of how much hemoglobin is saturated with oxygen
RDI (Respiratory disturbance index) | baseline
  Number of apneas, hypopneas and respiratory-effort related arousals (RERAs) per hour of sleep which is an indicator of severity of sleep apnea
Sleep/wake state | baseline
  Percentage of sleep and wake state
REM sleep | baseline
  Percentage of REM sleep
Deep sleep | baseline
  Percentage of deep sleep
Light sleep | baseline
  Percentage of light sleep
Sleep latency | baseline
  Latency of start of sleep in minutes
REM latency | baseline
  Latency of start of REM sleep in minutes
Total sleep time | baseline
  Total sleep time in minutes
Epworth sleepiness scale score (ESS) | at follow up after completion of treatment period (an average of three weeks)
  an 8-item questionnaire which takes about three minutes to fill out. It reflects the chance of each person's general level of sleepiness during eight situations of daily life. The subject selects the most appropriate integer score ranging from 0 (would never doze) to 3 (high chance of dozing) for each of the 8 questions. The results are then summed up, with 0 being the minimal and 24 the maximum total ESS score. The higher the ESS score, the higher that person's average sleep propensity in daily life. (0-5=Lower Normal Daytime Sleepiness, 6-10 = Higher Normal Daytime Sleepiness, 11-12 = Mild Excessive Daytime Sleepiness, 13-15 = Moderate Excessive Daytime Sleepiness, 16-24 =Severe Excessive Daytime Sleepiness.)
VAS (visual analogue scale) for snoring | at follow up after completion of treatment period (an average of three weeks)
  A standard 10-point VAS ranging from 0 (no snoring) to 10 (extreme snoring causing the bed partner to leave the bedroom or sleep separately) will be used to evaluate the subjective status of snoring during sleep. Heavy snoring corresponds to a snoring index of at least 7. A decrease of 3 points after treatment is considered significant. A satisfactory improvements is defined as a reduction to an index that is no longer experiences as bothersome (i.e. <3).
ODI (oxygen desaturation index) | at follow up after completion of treatment period (an average of three weeks)
  The ODI represents the average number of desaturation episodes (≥3%) per hour sleep.
PAT (peripheral arterial tone) signal | at follow up after completion of treatment period (an average of three weeks)
  PAT™ technology is a non-invasive window to the cardiovascular system and autonomic nervous system. Peripheral Arterial Tone (PAT™) signal is a proprietary technology used for non-invasively measuring arterial tone changes in peripheral arterial beds.
Heart rate | at follow up after completion of treatment period (an average of three weeks)
  The number of times a person's heart beats per minute. Normal heart rate range for adults is 60 to 100 beats per minute.
Body position | at follow up after completion of treatment period (an average of three weeks)
  Percentage of supine, prone, left, right, upright position
Snoring | at follow up after completion of treatment period (an average of three weeks)
  Snoring loudness in decibels
Oxygen saturation (SaO2) | at follow up after completion of treatment period (an average of three weeks)
  A measurement of the percentage of how much hemoglobin is saturated with oxygen
RDI (Respiratory disturbance index) | at follow up after completion of treatment period (an average of three weeks)
  Number of apneas, hypopneas and respiratory-effort related arousals (RERAs) per hour of sleep which is an indicator of severity of sleep apnea
Sleep/wake state | at follow up after completion of treatment period (an average of three weeks)
  Percentage of sleep and wake state
REM sleep | at follow up after completion of treatment period (an average of three weeks)
  Percentage of REM sleep
Deep sleep | at follow up after completion of treatment period (an average of three weeks)
  Percentage of deep sleep
Light sleep | at follow up after completion of treatment period (an average of three weeks)
  Percentage of light sleep
Sleep latency | at follow up after completion of treatment period (an average of three weeks)
  Latency of start of sleep in minutes
REM latency | at follow up after completion of treatment period (an average of three weeks)
  Latency of start of REM sleep in minutes
Total sleep time | at follow up after completion of treatment period (an average of three weeks)
  Total sleep time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Study Chair — Head of ENT department, UZA
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okuno K, Ono Minagi H, Ikai K, Matsumura Ai E, Takai E, Fukatsu H, Uchida Y, Sakai T. The efficacy of nasal airway stent (Nastent) on obstructive sleep apnoea and prediction of treatment outcomes. J Oral Rehabil. 2019 Jan;46(1):51-57. doi: 10.1111/joor.12725. Epub 2018 Oct 21. PMID 30281824
- [Background] Kumar AR, Guilleminault C, Certal V, Li D, Capasso R, Camacho M. Nasopharyngeal airway stenting devices for obstructive sleep apnoea: a systematic review and meta-analysis. J Laryngol Otol. 2015 Jan;129(1):2-10. doi: 10.1017/S0022215114003119. Epub 2014 Dec 29. PMID 25544266